CLINICAL TRIAL: NCT00736684
Title: Proximal Femoral Nail Antirotation™ (PFNA) Versus Gamma Nail 3™ (Gamma3) for Intramedullary Nailing of Unstable Trochanteric Fractures - a Multicenter Randomized Controlled Trial
Brief Title: Proximal Femoral Nail Antirotation™ (PFNA) Versus Gamma Nail 3™ (Gamma3) for Intramedullary Nailing of Unstable Trochanteric Fractures
Acronym: PROGAINT-ES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Collaborators: Synthes Inc. (Industry)
Responsible Party: Javier Vaquero Martin, MD, Hospital Gregorio Marañon
Organization: AO Innovation Translation Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROGAINT-ES-08
Record Dates: First submitted 2008-08-15; First posted 2008-08-18 (Estimated); Last update posted 2011-02-11 (Estimated); Status verified 2011-02

CONDITIONS: Unstable Trochanteric Fractures
Keywords: Femoral fractures [MeSH]; hip fractures [MeSH]; trochanteric fractures (femoral neck fractures [MeSH]); intramedullary nailing (fracture fixation, intramedullary [MeSH]); complex femoral fractures; femoral nail; surgical treatment (surgical procedures, operative [MeSH]); complications
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Proximal Femoral Nail AntirotationTM (PFNA)
  Interventions: Device: Proximal Femoral Nail AntirotationTM (PFNA)
- 2 (Other): Gamma Nail 3TM (Gamma3)
  Interventions: Device: Gamma Nail 3TM (Gamma3)

INTERVENTIONS:
Device: Proximal Femoral Nail AntirotationTM (PFNA) — intramedullary nailing
  Arms: 1
Device: Gamma Nail 3TM (Gamma3) — intramedullary nailing
  Arms: 2

SUMMARY:
The purpose of this study is to compare rates of any fracture fixation complication and revision rates after intramedullary fixation of unstable trochanteric fractures between the Proximal Femoral Nail Antirotation™ (PFNA)(Investigational Group) and Gamma Nail 3™ (Gamma3) (Control Group).

DETAILED DESCRIPTION:
Intramedullary nailing of unstable per- and subtrochanteric femoral fractures is a standard procedure in trauma and orthopaedic surgery. Unstable fractures treated with intramedullary nailing carry the risk of fracture fixation complications. The PFNA (Synthes) has evolved from the original PFN design, featuring a novel antirotation screw. Apart from the prevention of excess rotational forces, this supporting element may enhance the overall stability of the construct, thus potentially reducing fracture fixation complications. Empirical information about the fracture fixation complication rates of the PFNA device is not available. The primary objective of this study is to compare the 1-year fracture fixation rates between the PFNA and Gamma Nail 3™ (Stryker). Secondary objectives of the study are to compare differences in functional outcomes, quality of life outcomes, safety, radiological outcomes, handling and perceived effectiveness between the devices.

ELIGIBILITY:
Inclusion Criteria:

* Age 55 years and more
* Patients with isolated, unstable, closed or type 1 open trochanteric fractures, classified as AO 31-A2 or AO 31-A3
* Definitive primary fracture treatment with PFNA or Gamma3 (defined inTable 1) within three days after the index event
* Signed written informed consent (by the subjects or legal guardian) and agreement to attend the planned follow-ups

Exclusion Criteria:

* Pathologic fracture of any other cause than osteoporosis
* Patients or legal guardian refusing to sign the informed consent form
* Multiple trauma
* Type 2 and 3 open fractures
* Drug or alcohol abuse
* Wound and/or bone healing disorders of any other cause than diabetes mellitus or smoking
* Active malignancy
* Expected life expectancy ≤ 3 months
* Inability to walk independently prior to injury event (use of one stick is allowed. Not meeting inclusion criteria are bedridden, wheel-chair ridden and walker dependent subjects)
* Neurological and psychiatric disorders that would preclude reliable assessment (eg,, Parkinson disease, Multiple sclerosis, severe depression)
* Rheumatoid arthritis

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2007-11; Primary Completion 2009-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Any fracture fixation complication. | One year

SECONDARY OUTCOMES:
Bone union/fusion as evaluated by CT-scanning, health-related quality of life, disease-specific functional scoring, activities of daily living, mortality, radiological parameters, surgery details and surgeons' evaluation of handling and effectiveness. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Beate P. Hanson, MD, Study Director — AO Clinical Investigation and Documentation, Davos, Switzerland; Javier Vaquero Martin, MD, Principal Investigator — Hospital Gregorio Marañon, Madrid, Spain
Locations (6):
- Spain (6):
  - Hospital Universitario "Marqués de Valdecilla", Santander, Cantabria
  - Hospital Clinic, Barcelona, Catalonia
  - Hospital Gregorio Marañon, Madrid, Madrid
  - Hospital Puerta de Hierro, Madrid, Madrid
  - H.U. Virgen de la Arrixaca, Murcia
  - Hospital Donostia, San Sebastián